CLINICAL TRIAL: NCT07092475
Title: The Impact of Intraoperative Methadone on Postoperative Opioid Use
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study team will no longer be enrolling patients for this research.
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HCI182069
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Opioid Use
MeSH Terms: conditions — Breast Neoplasms | interventions — Amidines; Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The anesthesiology provider assigned to the patient's surgery will be notified of which treatment arm the patient is assigned to by the research coordinator or by the Director of Anesthesia Services on the day of surgery. The reconstructive surgeon and all other hospital staff (e.g. nurses) will be blinded to what treatment arm the patient was assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intraoperative Methadone (Experimental): the methadone group will receive a single dose of intravenous methadone administered within 30 minutes after induction of anesthesia by the attending anesthesiologist. The standard dose will be 20 mg, except for patients under 60 kg or over 65 years of age, who will receive 15 mg.
  Interventions: Drug: Methadon
- Control (No Intervention): The control group will not receive methadone and will instead receive a standard dose of 1 mg IV hydromorphone within the final 30-45 minutes of the procedure.

INTERVENTIONS:
Drug: Methadon — A long-acting synthetic opioid with a pharmacologic profile that potentially offers more stable and longer-lasting pain relief.
  Other Names: Diskets; Methadone Intensol; Methadose
  Arms: Intraoperative Methadone

SUMMARY:
This is a single-institution, randomized controlled trial to assess the effectiveness of intraoperative methadone on postoperative opioid use, pain control, and recovery in patients undergoing autologous breast reconstruction. Findings from this trial would inform subsequent perioperative pain protocols and allow the possible integration of intraoperative methadone into multimodal analgesia protocols.

DETAILED DESCRIPTION:
Opioid over prescription remains a significant contributor to the opioid crisis in the United States. One major contributor to this epidemic is postoperative opioid prescribing-over 80% of surgical patients receive opioids for postoperative pain, placing many, especially opioid-naive patients, at risk for prolonged use, dependence, and addiction.

Many traditional pain management interventions rely on high doses of short-acting opioids such as hydromorphone and fentanyl. Though effective in the short term, these medications often have fluctuating blood concentration levels, which can lead to ineffective pain control, increased side effects, and higher risk for long-term dependence and chronic use. Despite national efforts to promote better recovery pathways through multimodal pain management plans, significant variation in postoperative opioid prescribing and consumption patterns remains, and over 40% of surgical patients still do not achieve adequate relief of pain.

An alternative solution is intraoperative methadone, a long-acting synthetic opioid with a pharmacologic profile that potentially offers more stable and longer-lasting pain relief. Unlike short-acting opioids, a single dose of methadone given intraoperatively has been shown to be capable of maintaining analgesic levels for up to 24-36 hours, potentially reducing total postoperative opioid requirements.

The use of intraoperative methadone for cardiac, spine, and ambulatory procedures is well-established, demonstrating that methadone leads to significant reductions in perioperative opioid use and pain scores postoperatively without increased risk of opioid side effects. In addition, preliminary data from a 2022 study on DIEP flap patients and a 2024 retrospective cohort study on mastectomy patients both suggest that intraoperative methadone significantly reduces postoperative opioid requirements.

Preliminary retrospective data from revealed that patients receiving intraoperative methadone for autologous breast reconstruction had significantly lower postoperative opioid consumption compared to those who did not receive intraoperative methadone, with a 37.2% reduction in total inpatient opioid use. However, prospective, randomized data in this population is currently lacking.

This is a single-institution, randomized controlled trial to assess the effectiveness of intraoperative methadone on postoperative opioid use, pain control, and recovery in patients undergoing autologous breast reconstruction. Findings from this trial would inform subsequent perioperative pain protocols and allow the possible integration of intraoperative methadone into multimodal analgesia protocols.

Patients will be randomized to either a methadone cohort or a control cohort. Aside from this intervention, both groups will undergo the same standardized intraoperative anesthetic protocol. Surgical care will not be altered for study purposes.

Postoperative care will follow institutional protocols and will not be altered for study purposes. Patients in both cohorts will receive the same standardized postoperative analgesic regimen, including as-needed (PRN) administration of short-acting opioids (e.g., IV hydromorphone, IV fentanyl), acetaminophen, and antiemetics. NSAIDs such as ketorolac or celecoxib will be avoided.

Patients will be monitored daily for opioid-related side effects including nausea, vomiting, constipation, sedation, and respiratory depression. Nausea will be assessed both through direct patient report and review of antiemetic administration (e.g., ondansetron, metoclopramide).

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Patients undergoing unilateral or bilateral autologous breast reconstruction with abdominally-based free flaps after mastectomy for breast cancer or cancer prophylaxis

Exclusion Criteria:

* Patients undergoing reoperations such as autologous breast reconstruction as a revision procedure following failed implant-based reconstruction
* Patients undergoing multiple procedures such as mastectomy and immediate reconstruction
* Patients with documented chronic opioid use prior to procedure, or chronic pain condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Total Postoperative Opioid Use | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  Total perioperative opioid consumption will be measured in morphine milligram equivalents (MMEs), a standardized measure to quantify the strength of opioid doses compared to morphine.
  This outcome measure will be assessed from the day of surgery until discharge, up to 4 weeks.

SECONDARY OUTCOMES:
Patient-Reported Pain Scores - Visual Analog Scale | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  This outcome measure will assess visual analog scale scores, a measurement to assess pain by having subjects mark pain on a line. Visual analog scale scores range from 0-10, with lower scores indicating less perceived pain and higher scores indicating more perceived pain.
Patient-Reported Pain Scores - Pain Interference Score | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  This outcome measure will assess pain interference scores, a measure for assessing how pain impacts daily life.
  Pain Interference scores range from 0-10, with lower scores indicating less interference with daily life and higher scores indicating more interference with daily life.
Patient-Reported Pain Scores - Patient Pain Management Satisfaction Scale | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  This outcome measure will assess patient pain management satisfaction scale scores in the immediate postoperative period.
  The Patient Pain Management Satisfaction Scale is a single-item, self-reported question, "Please write your satisfaction with your pain management". Patient Pain Management Satisfaction Scale scores range from 0 to 100, with lower scores indicating worse satisfaction with pain management and higher scores indicating better satisfaction with pain management.
Length of hospital stay | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  Length of hospital stay will be captured in 24-hour intervals. This outcome measure will report the mean hospital stay in days.
Proportion of participants utilizing non-opioid analgesics | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  This outcome measure will report the proportion of participants who used non-opioid analgesics such as Tylenol (Acetaminophen) and NSAIDs.
Days of non-opioid analgesics use | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  This outcome measure will report the mean days research participants took non-opioid analgesics.
Opioid-related side effects | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  Patients will be monitored daily for opioid-related side effects, including nausea, vomiting, constipation, sedation, and respiratory depression. This outcome measure will report the proportion of subjects who experience each opioid-related side effect.
Time to opioid cessation | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  This outcome measure will report the mean time in days to opioid cessation for each group.
Complication Rates | from the day of surgery until discharge, up to 4 weeks.
  To evaluate the impact of intraoperative methadone administration on postoperative opioid use and pain control in patients undergoing autologous breast reconstruction.
  Patients will be monitored daily for surgery complications, including wound issues, seroma/hematoma, infection, takeback to OR, readmission, ED visits, and reoperation. This outcome measure will report the proportion of subjects who experience each complications.

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Kwok, MD, MPH, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Joy Ha, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CfDCa Prevention: Opioids. https://www.cdc.gov/opioids/index.html. Accessed October 26, 2021.
- [Background] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Background] Olds C, Spataro E, Li K, Kandathil C, Most SP. Assessment of Persistent and Prolonged Postoperative Opioid Use Among Patients Undergoing Plastic and Reconstructive Surgery. JAMA Facial Plast Surg. 2019 Jul 1;21(4):286-291. doi: 10.1001/jamafacial.2018.2035. PMID 30844024
- [Background] Mercadante S. Intravenous Methadone for Perioperative and Chronic Cancer Pain: A Review of the Literature. Drugs. 2023 Jul;83(10):865-871. doi: 10.1007/s40265-023-01876-7. Epub 2023 Jun 13. PMID 37308798
- [Background] Barker JC, DiBartola K, Wee C, Andonian N, Abdel-Rasoul M, Lowery D, Janis JE. Preoperative Multimodal Analgesia Decreases Postanesthesia Care Unit Narcotic Use and Pain Scores in Outpatient Breast Surgery. Plast Reconstr Surg. 2018 Oct;142(4):443e-450e. doi: 10.1097/PRS.0000000000004804. PMID 29979365
- [Background] Muetterties CE, Taylor JM, Kaeding DE, Morales RR, Nguyen AV, Kwan L, Tseng CY, Delong MR, Festekjian JH. Enhanced Recovery after Surgery Protocol Decreases Length of Stay and Postoperative Narcotic Use in Microvascular Breast Reconstruction. Plast Reconstr Surg Glob Open. 2023 Dec 14;11(12):e5444. doi: 10.1097/GOX.0000000000005444. eCollection 2023 Dec. PMID 38098953
- [Background] Gort N, van Gaal BGI, Tielemans HJP, Ulrich DJO, Hummelink S. Positive effects of the enhanced recovery after surgery (ERAS) protocol in DIEP flap breast reconstruction. Breast. 2021 Dec;60:53-57. doi: 10.1016/j.breast.2021.08.010. Epub 2021 Aug 20. PMID 34464847
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Kharasch ED, Brunt LM, Blood J, Komen H. Intraoperative Methadone in Next-day Discharge Outpatient Surgery: A Randomized, Double-blinded, Dose-finding Pilot Study. Anesthesiology. 2023 Oct 1;139(4):405-419. doi: 10.1097/ALN.0000000000004663. PMID 37350677
- [Background] Udelsmann A, Maciel FG, Servian DC, Reis E, de Azevedo TM, Melo Mde S. Methadone and morphine during anesthesia induction for cardiac surgery. Repercussion in postoperative analgesia and prevalence of nausea and vomiting. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):695-701. doi: 10.1016/S0034-7094(11)70078-2. English, Multiple languages. PMID 22063370
- [Background] Carle N, Nikolajsen L, Uhrbrand CG. Respiratory Depression Following Intraoperative Methadone: A Retrospective Cohort Study. Anesth Analg. 2025 Mar 1;140(3):516-523. doi: 10.1213/ANE.0000000000007018. Epub 2025 Feb 14. PMID 38814334
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Vender JS, Benson J, Newmark RL. Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Posterior Spinal Fusion Surgery: A Randomized, Double-blinded, Controlled Trial. Anesthesiology. 2017 May;126(5):822-833. doi: 10.1097/ALN.0000000000001609. PMID 28418966
- [Background] Bernstein JL, Lu Wang M, Huang H, Otterburn DM. Intra-operative Methadone Decreases Post-operative Pain and Opioid Use in DIEP Flap Breast Patients: A New ERAS Protocol. Plast Reconstr Surg Glob Open. 2022;10(10 Suppl):92. Published 2022 Oct 24. doi:10.1097/01.GOX.0000898792.35273.f6
- [Background] NIDA. Drug Overdose Deaths: Facts and Figures. National Institute on Drug Abuse website. https://nida.nih.gov/research-topics/trends-statistics/overdose-death-rates. August 21, 2024 Accessed November 12, 2024.
- [Background] Centers for Disease Control and Prevention. State Unintentional Drug Overdose Reporting System (SUDORS). Preliminary Data. Atlanta, GA: US Department of Health and Human Services, CDC; November 12, 2024. Access at: https://www.cdc.gov/overdose-prevention/data-research/facts-stats/sudors-dashboard-fatal-overdose-data.html
- [Background] Florence C, Luo F, Rice K. The economic burden of opioid use disorder and fatal opioid overdose in the United States, 2017. Drug Alcohol Depend. 2021 Jan 1;218:108350. doi: 10.1016/j.drugalcdep.2020.108350. Epub 2020 Oct 27. PMID 33121867
- [Background] Meyer R, Patel AM, Rattana SK, Quock TP, Mody SH. Prescription opioid abuse: a literature review of the clinical and economic burden in the United States. Popul Health Manag. 2014 Dec;17(6):372-87. doi: 10.1089/pop.2013.0098. PMID 25075734
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Alam A, Gomes T, Zheng H, Mamdani MM, Juurlink DN, Bell CM. Long-term analgesic use after low-risk surgery: a retrospective cohort study. Arch Intern Med. 2012 Mar 12;172(5):425-30. doi: 10.1001/archinternmed.2011.1827. PMID 22412106
- [Background] Goldberg RF. The Opioid Crisis: The Surgeon's Role. Adv Surg. 2019 Sep;53:305-325. doi: 10.1016/j.yasu.2019.04.015. Epub 2019 May 17. No abstract available. PMID 31327454
- [Background] Theisen K, Jacobs B, Macleod L, Davies B. The United States opioid epidemic: a review of the surgeon's contribution to it and health policy initiatives. BJU Int. 2018 Nov;122(5):754-759. doi: 10.1111/bju.14446. Epub 2018 Jul 26. PMID 29896932
- [Background] Murphy GS, Szokol JW. Intraoperative Methadone in Surgical Patients: A Review of Clinical Investigations. Anesthesiology. 2019 Sep;131(3):678-692. doi: 10.1097/ALN.0000000000002755. No abstract available. PMID 31094758
- [Background] Lai G, Aroke EN, Zhang SJ. Rediscovery of Methadone to Improve Outcomes in Pain Management. J Perianesth Nurs. 2022 Aug;37(4):425-434. doi: 10.1016/j.jopan.2021.08.011. Epub 2022 Apr 6. PMID 35396188
- [Background] Temple-Oberle C, Shea-Budgell MA, Tan M, Semple JL, Schrag C, Barreto M, Blondeel P, Hamming J, Dayan J, Ljungqvist O; ERAS Society. Consensus Review of Optimal Perioperative Care in Breast Reconstruction: Enhanced Recovery after Surgery (ERAS) Society Recommendations. Plast Reconstr Surg. 2017 May;139(5):1056e-1071e. doi: 10.1097/PRS.0000000000003242. PMID 28445352
- [Background] Jablonka EM, Lamelas AM, Kim JN, Molina B, Molina N, Okwali M, Samson W, Sultan MR, Dayan JH, Smith ML. Transversus Abdominis Plane Blocks with Single-Dose Liposomal Bupivacaine in Conjunction with a Nonnarcotic Pain Regimen Help Reduce Length of Stay following Abdominally Based Microsurgical Breast Reconstruction. Plast Reconstr Surg. 2017 Aug;140(2):240-251. doi: 10.1097/PRS.0000000000003508. PMID 28746269
- [Background] Carron M, Tamburini E, Linassi F, Pettenuzzo T, Boscolo A, Navalesi P. Efficacy of nonopioid analgesics and adjuvants in multimodal analgesia for reducing postoperative opioid consumption and complications in obesity: a systematic review and network meta-analysis. Br J Anaesth. 2024 Dec;133(6):1234-1249. doi: 10.1016/j.bja.2024.08.009. Epub 2024 Oct 3. PMID 39366846
- [Background] Tageza Ilala T, Teku Ayano G, Ahmed Kedir Y, Tamiru Mamo S. Evidence-Based Guideline on the Prevention and Management of Perioperative Pain for Breast Cancer Peoples in a Low-Resource Setting: A Systematic Review Article. Anesthesiol Res Pract. 2023 Nov 3;2023:5668399. doi: 10.1155/2023/5668399. eCollection 2023. PMID 37953883
- [Background] Baratta JL, Schwenk ES, Viscusi ER. Clinical consequences of inadequate pain relief: barriers to optimal pain management. Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):15S-21S. doi: 10.1097/PRS.0000000000000681. PMID 25254999
- [Background] Lawal OD, Gold J, Murthy A, Ruchi R, Bavry E, Hume AL, Lewkowitz AK, Brothers T, Wen X. Rate and Risk Factors Associated With Prolonged Opioid Use After Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jun 1;3(6):e207367. doi: 10.1001/jamanetworkopen.2020.7367. PMID 32584407
- [Background] Glowacki D. Effective pain management and improvements in patients' outcomes and satisfaction. Crit Care Nurse. 2015 Jun;35(3):33-41; quiz 43. doi: 10.4037/ccn2015440. PMID 26033099
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331
- [Background] Sunilkumar MM, Lockman K. Practical Pharmacology of Methadone: A Long-acting Opioid. Indian J Palliat Care. 2018 Jan;24(Suppl 1):S10-S14. doi: 10.4103/IJPC.IJPC_180_17. PMID 29497249
- [Background] Hanna V, Senderovich H. Methadone in Pain Management: A Systematic Review. J Pain. 2021 Mar;22(3):233-245. doi: 10.1016/j.jpain.2020.04.004. Epub 2020 Jun 26. PMID 32599153
- [Background] Komen H, Brunt LM, Deych E, Blood J, Kharasch ED. Intraoperative Methadone in Same-Day Ambulatory Surgery: A Randomized, Double-Blinded, Dose-Finding Pilot Study. Anesth Analg. 2019 Apr;128(4):802-810. doi: 10.1213/ANE.0000000000003464. PMID 29847382
- [Background] Broyles JM, Balk EM, Adam GP, Cao W, Bhuma MR, Mehta S, Dominici LS, Pusic AL, Saldanha IJ. Implant-based versus Autologous Reconstruction after Mastectomy for Breast Cancer: A Systematic Review and Meta-analysis. Plast Reconstr Surg Glob Open. 2022 Mar 11;10(3):e4180. doi: 10.1097/GOX.0000000000004180. eCollection 2022 Mar. PMID 35291333
- [Background] Jacobs A, Lemoine A, Joshi GP, Van de Velde M, Bonnet F; PROSPECT Working Group collaborators#. PROSPECT guideline for oncological breast surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2020 May;75(5):664-673. doi: 10.1111/anae.14964. Epub 2020 Jan 26. PMID 31984479
- [Background] Roth RS, Lowery JC, Davis J, Wilkins EG. Persistent pain following postmastectomy breast reconstruction: long-term effects of type and timing of surgery. Ann Plast Surg. 2007 Apr;58(4):371-6. doi: 10.1097/01.sap.0000239810.38137.84. PMID 17413877
- [Background] Cata JP, Zaidi Y, Guerra-Londono JJ, Kharasch ED, Piotrowski M, Kee S, Cortes-Mejia NA, Gloria-Escobar JM, Thall PF, Lin R. Intraoperative methadone administration for total mastectomy: A single center retrospective study. J Clin Anesth. 2024 Nov;98:111572. doi: 10.1016/j.jclinane.2024.111572. Epub 2024 Aug 23. PMID 39180867
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Gordon DB, Dahl JL, Miaskowski C, McCarberg B, Todd KH, Paice JA, Lipman AG, Bookbinder M, Sanders SH, Turk DC, Carr DB. American pain society recommendations for improving the quality of acute and cancer pain management: American Pain Society Quality of Care Task Force. Arch Intern Med. 2005 Jul 25;165(14):1574-80. doi: 10.1001/archinte.165.14.1574. PMID 16043674
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683